CLINICAL TRIAL: NCT02583750
Title: Snooze Control: The Effect of Sleep Deprivation on Glucose Metabolism
Brief Title: Snooze Control: Sleep Duration & Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuewen Wang (Other)
Responsible Party: Sponsor-Investigator, Xuewen Wang, Dr. Xuewen Wang, PhD., University of South Carolina
Organization: University of South Carolina (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00032421
Record Dates: First submitted 2015-10-15; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Glucose Metabolism Disorders
Keywords: glucose metabolism; sleep deprivation
MeSH Terms: conditions — Glucose Metabolism Disorders; Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OGTT after deprived sleep first (Experimental): Participants came to the lab to perform the oral glucose tolerance test after three nights of sleep deprivation, then another test after three nights of sufficient sleep
  Interventions: Behavioral: OGTT after deprived sleep first
- OGTT after sufficient sleep first (Experimental): Participants came to the lab to perform the oral glucose tolerance test after three nights of sufficient sleep, then another test after three nights of deprived sleep
  Interventions: Behavioral: OGTT after sufficient sleep first

INTERVENTIONS:
Behavioral: OGTT after deprived sleep first — Participants slept 1-3 hours less than their normal amount for three nights, and then came to the lab for the oral glucose tolerance testing after a 12 hour overnight fast. The second oral glucose tolerance test was after they slept as much as they wanted for three nights.
  Arms: OGTT after deprived sleep first
Behavioral: OGTT after sufficient sleep first — Participants slept as much as they wanted for three nights, and then came to the lab for the oral glucose tolerance testing after a 12 hour overnight fast. The second oral glucose tolerance test was after they slept 1-3 hours less than normal for three nights.
  Arms: OGTT after sufficient sleep first

SUMMARY:
This project investigated how glucose metabolism differs due to sleep deprivation for three consecutive nights as compared to sufficient sleep for three nights by examining concentrations of glucose, insulin, and other factors involved in glucose metabolism.

DETAILED DESCRIPTION:
16 participants were enrolled in the study (8 females, 8 males) aged 18-25 years. In order for the participants to qualify for the study, each had to wear a pedometer for a week before the study began to determine eligibility. Each participant came to the lab for an oral glucose tolerance test on a morning, following three nights when they were sleep deprived, and on another morning when they had three nights' sufficient sleep. The sequence of the oral glucose tolerance tests were randomly assigned. The sleep duration for participants was monitored by the readings of the sleep monitors that each participant wore. The oral glucose tolerance tests were performed after an overnight fast. A 20-gauge polyethylene catheter was placed in the antecubital vein for blood sampling. Blood samples were drawn once (0 min) before and 4 times (30, 60, 90, and 120 min) after a 75g glucose drink was consumed for the determination of plasma glucose, insulin, and concentrations of other factors. Each participant was told to continue their regular routine during the study period, including diet, caffeine usage, and exercise.

ELIGIBILITY:
Inclusion Criteria:

* healthy college-aged males and females
* being minimally active

Exclusion Criteria:

* average more than 15,000 steps a day
* major health issues such as heart disease, diabetes
* taking medication to help with sleep or using a sleeping device
* any type of sleep problem such as sleep apnea

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Glucose concentrations during oral glucose tolerance test | two hours

CONTACTS AND LOCATIONS:
Overall Officials: Xuewen Wang, PhD, Principal Investigator — University of South Carolina
Locations (1):
- Public Health Research Center University of South Carolina, Columbia, South Carolina, United States